CLINICAL TRIAL: NCT05701059
Title: Comparison of Unconstrained and Semi-constrained Artificial Disc Implants Used in Cervical Disc Arthroplasty
Brief Title: Comparison of Artificial Disc Implants in Cervical Disc Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Principal Investigator, Neuroplasticity and Repair Laboratory, University of California, Los Angeles
Other Study IDs: 22-001808
Record Dates: First submitted 2022-12-13; First posted 2023-01-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cervical Spondylosis with Myelopathy; Cervical Radiculopathy; Cervical Disc Herniation; Degenerative Disc Disease
Keywords: cervical; spondylosis; myelopathy; radiculopathy; disc; cervical disc; artificial disc; artificial disc implantation; cervical arthroplasty; disc herniation; degenerative disc disease; ACDF; Biomet Zimmer Mobi-C; Nuvasive Simplify
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Degeneration; Spondylosis; Spinal Cord Diseases; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Semi-Constrained Nuvasive Simplify: This group will be undergoing cervical arthroplasty with the Nuvasive Simplify artificial disc implant. The Nuvasive Simplify implements a three-piece design with two endplates and a semi-constrained mobile core.
  Interventions: Procedure: Cervical arthroplasty; Device: Semi-Constrained Nuvasive Simplify
- Unconstrained Biomet Zimmer Mobi-C: This group will be undergoing cervical arthroplasty with the Biomet Zimmer Mobi-C artificial disc implant. The Biomet Zimmer Mobi-C implements an unconstrained three piece design.
  Interventions: Procedure: Cervical arthroplasty; Device: Unconstrained Biomet Zimmer Mobi-C

INTERVENTIONS:
Procedure: Cervical arthroplasty — A joint replacement procedure administered by inserting an artificial disc between the vertebrae to replace a natural spinal disc after it has been removed.
  Other Names: Cervical artificial disc replacement surgery
Device: Semi-Constrained Nuvasive Simplify — This weight-bearing implant consisting of PEEK (polyetheretherketone) endplates and one semi-constrained, fully articulating, mobile zirconia toughened alumina (ZTA) ceramic core will be administered by cervical arthroplasty into the specified single-level cervical region.
  Groups: Semi-Constrained Nuvasive Simplify
Device: Unconstrained Biomet Zimmer Mobi-C — This unconstrained, three-piece implant will be administered by cervical arthroplasty into the specified single-level cervical region.
  Groups: Unconstrained Biomet Zimmer Mobi-C

SUMMARY:
This study will comprehensively evaluate the outcomes and endpoints of these two different FDA-approved artificial disc implants used to treat cervical spondylotic myelopathy and/or radiculopathy today: Biomet Zimmer Mobi-C and Nuvasive Simplify. Both implants are structurally different with the Nuvasive Simplify implementing a three-piece design with two endplates and a semi-constrained mobile core while the Biomet Zimmer Mobi-C implements an unconstrained three piece design. Subjects will be age-matched and randomly assigned to either implant with informed consent. All subjects will undergo a variety of assessments that evaluate neck disability, quality of life, pain, physiological outcome (radiographic assessments), and neck range-of motion before and after their procedure. One baseline testing will be conducted along with three post-operation visits (three months, six months, and one year) in accordance to standard follow-up procedure. Thus, the duration of participation in the study will be approximately one and a half years.

DETAILED DESCRIPTION:
In cases where surgery is indicated, treatment for cervical spondylotic myelopathy and/or radiculopathy (typically caused by disc herniation or degenerative disc disease) has traditionally been performed by a procedure known as anterior cervical discectomy and fusion (ACDF) to treat a damaged disc in the neck area of the spine. However, medical advancement in this field has allowed for a new procedure often referred to as cervical arthroplasty that implements artificial disc implantation. These implants mimic the function and structure of discs by cushioning the neck's vertebral bones instead of fusing them and providing flexibility for head movements. The emergence of different artificial disc implants that are structurally and mechanistically different calls for a comparative analysis that evaluates performance across a comprehensive set of patient outcomes.

This study will comprehensively evaluate the outcomes and endpoints of these two different FDA-approved artificial disc implants used to treat cervical spondylotic myelopathy and/or radiculopathy today: Biomet Zimmer Mobi-C and Nuvasive Simplify. Both implants are structurally different with the Nuvasive Simplify implementing a three-piece design with two endplates and a semi-constrained mobile core while the Biomet Zimmer Mobi-C implements an unconstrained three piece design. Subjects will be age-matched and randomly assigned to either implant with informed consent. All subjects will undergo a variety of assessments that evaluate neck disability, quality of life, pain, physiological outcome (radiographic assessments), and neck range-of motion before and after their procedure. One baseline testing will be conducted along with three post-operation visits (three months, six months, and one year) in accordance to standard follow-up procedure. Thus, the duration of participation in the study will be approximately one and a half years.

This study has significant implications in better assessing the overall efficacy of cervical arthroplasty while providing insight to the differences in outcomes based on the artificial disc implanted. Findings can also contribute to characterizing the advantages and disadvantages of both implants to aid surgeons in making more informed and personalized treatment recommendations according to the needs of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature and between 18 to 60 years of age
* Experiences cervical spondylotic myelopathy and/or radiculopathy typically caused by disc herniation or degenerative disc disease at a single level between C3 to C7
* Is unresponsive to at least six weeks of non-surgical conservative care
* Has the intention of undergoing cervical arthroplasty for their chief complaint
* Signed informed consent form

Exclusion Criteria:

* Patient has had prior cervical spine surgery
* Has more than two diseased levels requiring surgery
* Has a known allergy to a metal alloy or polyethylene
* Is morbidly obese
* Has active local or system infection
* Has any circumstances or conditions such that their ability to provide informed consent comply with follow-up requirements, or provide self-assessments is compromised (eg: psychiatric disorders, chronic alcohol or substance abuse, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects must be experiencing cervical spondylotic myelopathy and/or radiculopathy typically caused by disc herniation or degenerative disc disease at a single level between C3 to C7 after being unresponsive to at least six weeks of non-surgical conservative care. This study is for patients who have the intention of undergoing cervical arthroplasty and have already been recommended to do so by a doctor.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cervical range of motion assessments with VICON | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Will measure flexion/extension, lateral bending, rotation, protraction/retraction in degrees. The outcome will reflect any improvement in physiological neck range of motion be patients undergoing this procedure.

SECONDARY OUTCOMES:
Questionnaires on neck disability | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Will administer surveys on neck disability index, work status, pain intensity worksheet, treatment satisfaction form, and the SF-12 v2 Health Survey. The 12-item Short Form Survey version 2 (SF-12 v2) is a general health questionnaire that reports two summary scores - a mental component score (MCS-12) and a physical component score (PCS-12). The scores are reported as Z-scores (difference compared to the population average, measured in standard deviations) with the US population average PCS-12 and MCS-12 being both 50 points. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. Overall, these assessments will help to gauge overall quality of life, pain, and patient satisfaction with their treatment.
Neurological examination: gait assessment | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Will take place as part of standard care for this operation. A gait assessment will be performed according to Nurick's Classification. Nurick's classification is graded from 0-5 or normal, with a number grade denoting some neurological deficit. 0 is least severe, with the patient showing root signs and symptoms with no evidence of spinal cord involvement. Grade 5 is most severe, described as chair bound or bedridden.
Neurological examination: foraminal compression test | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  The foraminal compression test is a physical examination technique which reduces the opening of the foramen which may demonstrate if there is pressure upon the exiting spinal nerve. The test is done to detect spinal nerve root involvement, a herniated disc, bulging disc, or foraminal stenosis. The scoring is binary, either negative or positive, to test for any pain the patient experiences during the exam.
Radiographic assessments: disc height | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Will take place as part of standard care for this operation. Anterior and Posterior Disc Height will be measured from neutral lateral radiographs. Anterior (Posterior) Disc Height is defined as the distance between the anterior-inferior (posterior-inferior) corner of the superior vertebra, and the corresponding corner of the inferior vertebra. This distance is measured perpendicular to the superior endplate of the inferior vertebra and will be reported in units of millimeters. Average Disc Height is calculated as the simple average of the Anterior and Posterior Disc Heights.
Radiographic assessments: disc angle | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Disc Angle is the angle formed between the endplates of adjacent vertebrae. Disc Angle will be measured on neutral lateral radiographs to assess local segmental lordosis and will be reported in degrees.
Radiographic assessments: global range of motion (C2-C6) | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Global range of motion will be measured on lateral flexion-extension views to evaluate global range of motion. Global C2-C6 range of motion will be calculated by subtracting the C2-C6 angle in flexion from the C2-C6 angle in extension. Global range of motion will be measured between the inferior endplate of C2 and the inferior endplate of C6. C2-C6 Angle will be measured in units of degrees.
Radiographic assessments: translational motion | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Translational Motion will be calculated from flexion-extension radiographs. Translational Motion is defined as displacement of the posterior-inferior corner of the superior vertebra in a direction defined parallel to the superior endplate of the inferior vertebra. Translational Motion will be reported in units of millimeters and as a percent of the AP dimension of the superior endplate of the inferior vertebra.
Radiographic assessments: device subsidence | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Device Subsidence will assess significant cranial-caudal movement of the implant and will be graded in accordance with the following definitions:
  0. None: No evidence of cranial or caudal subsidence of the implant > 3 mm.
  1. Cranial: Presence of cranial movement of the device > 3 mm relative to the initial position of the implant at PostOp.
  2. Caudal: Presence of caudal movement of the device > 3 mm relative to the initial position of the implant at PostOp.
  Subsidence will be evaluated relative to the first available post-operative visit. A threshold of >3 mm of implant motion will be used to define significance. Subsidence will be assessed in the cranial and caudal directions perpendicular to the vertebral endplates and based on the degree of penetration of the implant into the bony margins of the vertebral body.
Radiographic assessments: Kellgren-Lawrence Assessment | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Kellgren-Lawrence ALDD at the adjacent levels will be graded in accordance with the following definitions adapted from Kellgren and Lawrence:
  0. None: No degenerative changes.
  1. Doubtful: Minimal osteophytosis only.
  2. Minimal: Definite osteophytosis with some sclerosis of anterior part of vertebral plates.
  3. Moderate: Marked osteophytosis and sclerosis of vertebral plates with slight narrowing of disk space.
  4. Severe: Large osteophytes, marked sclerosis of vertebral plates, and marked narrowing of disk space.
  The assessment of Kellgren-Lawrence Osteoarthritis Grade will be graded by the reviewers based on an assessment from X-ray of three component factors: disc space narrowing (assessed relative to an nearby normal disc), osteophyte formation and endplate sclerosis.
Radiographic assessments: intervertebral angle (index and adjacent levels) | Will be conducted before surgery (baseline), and 3 months, 6 months, and 1 year post-operation.
  Intervertebral Angle is used to define the endplate angle of the superior vertebra relative to the inferior vertebra. The difference in the angles measured is equivalent to a change in the Disc Angle. Intervertebral Angles will be measured in the sagittal plane from flexion and extension images separately and in the coronal plane from left and right bending images separately. All values will be reported in degrees. Intervertebral Angle will be calculated from lateral flexion-extension radiographs. Intervertebral Angle, also known as rotation, is defined as the change in angle between the adjacent endplates of the motion segment. Intervertebral Angle will be reported in units of degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Lu, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No